CLINICAL TRIAL: NCT03280719
Title: Whole Breast (WB) + Lymph Node Irradiation (LNI): Prone Compared to Supine Position in a Randomized Study with 15 or 5 Fractions
Brief Title: Whole Breast + Lymph Node Irradiation: Prone Compared to Supine Position in 15 or 5 Fractions
Acronym: PRO-SURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/0256; CIV-BE-17-06-020245 (Other: EUDAMED)
Record Dates: First submitted 2017-08-02; First posted 2017-09-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasms; Radiotherapy; Lymph Node Metastases
Keywords: Prone position; Supine position; Hypofractionation; Accelerated radiotherapy; Regional nodal irradiation
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis; Deception | interventions — Acceleration; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Supine Hypofractionated Radiotherapy (Active Comparator): Supine Radiotherapy and Hypofractionation:
  Whole breast + regional nodal irradiation in supine position with a median dose of 15 x 2.67 Gy prescribed to the whole breast and nodal regions. Median dose of the simultaneously integrated boost is 3.12 Gy per fraction.
  Interventions: Device: Supine Radiotherapy; Radiation: Hypofractionation
- Prone Hypofractionated Radiotherapy (Experimental): Prone Radiotherapy and Hypofractionation:
  Whole breast + regional nodal irradiation in prone position with a 15 x 2.67 Gy dose prescription to the whole breast and nodal regions. Median dose of the simultaneously integrated boost is 3.12 Gy per fraction.
  Interventions: Device: Prone Radiotherapy; Radiation: Hypofractionation
- Supine Accelerated Radiotherapy (Experimental): Supine Radiotherapy and Acceleration:
  Whole breast + regional nodal irradiation in supine position with a median dose of 5 x 5.7 Gy to the whole breast. Lymph node regions receive a median dose of 5 x 5.4 Gy. Median dose of the simultaneously integrated boost is 6.2 Gy per fraction.
  Interventions: Radiation: Acceleration; Device: Supine Radiotherapy
- Prone Accelerated Radiotherapy (Experimental): Prone Radiotherapy and Acceleration:
  Whole breast + regional nodal irradiation in prone position with a median dose of 5 x 5.7 Gy to the whole breast. Lymph node regions receive a median dose of 5 x 5.4 Gy. Median dose of the simultaneously integrated boost is 6.2 Gy per fraction.
  Interventions: Device: Prone Radiotherapy; Radiation: Acceleration

INTERVENTIONS:
Device: Prone Radiotherapy — Prone positioning for regional nodal irradiation using the crawl breast couch.
  Other Names: Crawl position; Prone regional nodal irradiation
  Arms: Prone Accelerated Radiotherapy; Prone Hypofractionated Radiotherapy
Radiation: Acceleration — Accelerated irradiation in 5 fractions over 12 days with simultaneously integrated boost
  Other Names: HAI-5; Hyper-accelerated irradiation; 5 fractions
  Arms: Prone Accelerated Radiotherapy; Supine Accelerated Radiotherapy
Device: Supine Radiotherapy — Supine positioning for regional nodal irradiation using breastboard.
  Other Names: Supine regional nodal irradiation
  Arms: Supine Accelerated Radiotherapy; Supine Hypofractionated Radiotherapy
Radiation: Hypofractionation — Moderate hypofractionation in 15 fractions over 3 weeks with simultaneously integrated boost
  Other Names: Moderate hypofractionation
  Arms: Prone Hypofractionated Radiotherapy; Supine Hypofractionated Radiotherapy

SUMMARY:
The goal of this trial is to evaluate the effect of the prone crawl treatment position and/or accelerated schedule on acute and late toxicities, as well as quality of life and time management for breast cancer patients receiving whole breast and regional nodal irradiation after breast conserving surgery.

DETAILED DESCRIPTION:
Locoregional radiotherapy after lumpectomy and axillary node dissection diminishes the locoregional recurrence risk at 10 years by 21,2 % in women with pathologically confirmed lymph node involvement.

Excess dose to organs at risk can lead to acute and late side effects, such as tissue damage, organ malfunction and secondary cancers. Radiotherapy in prone position has helped reduce these risks for whole breast radiotherapy only, but has not yet been adequately investigated for patients also requiring regional nodal irradiation. One of the reasons is that there is no optimal patient support device available to allow regional nodal irradiation in prone position. To this end, a novel positioning device was developed at our center, allowing regional nodal irradiation in prone position. It was called the crawl breast couch because the patient position resembles a phase from the crawl swimming technique. A previous planning study by Deseyne et al. using this device shows a benefit (i.e. reduced dose) for the ipsilateral lung, the thyroid, as well as a minor benefit for the right lung, and contralateral breast (which already receive very low relative doses) while maintaining similar target coverage when compared to supine positioning.

Apart from the paradigm shift from supine to prone radiotherapy, in recent years, it has become clear that breast cancer cells are more sensitive to fraction dose than originally presumed. Large randomized trials confirm this hypothesis: moderate hypofractionation schemes in 15 or 16 fractions are at least equivalent in tumor control and toxicity although the total dose is lower than the traditional 50 Gy in 25 fractions. Further acceleration to 5 fractions is expected to have an even larger radiobiological advantage regarding tumor control. Additional advantages are patient comfort and a better use of radiotherapy resources.

This randomized trial with 2 x 2 factorial design tests 2 interventions for patients with breast cancer requiring whole-breast and regional nodal irradiation: radiotherapy in prone position with a specifically designed patient support device called the crawl breast couch, and accelerated radiotherapy in 5 fractions. The standard arm in this trial is supine hypofractionated radiotherapy.

The goal of this trial is to evaluate the effect of the prone crawl treatment position and/or accelerated schedule on acute and late toxicities, as well as quality of life and time management for breast cancer patients receiving whole breast and regional nodal irradiation after breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Breast conserving surgery
* AND Multidisciplinary decision of adjuvant whole breast + regional nodal irradiation
* AND Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* Mastectomy
* OR Bilateral breast irradiation
* OR Distant metastasis/metastases
* OR previous irradiation to the thoracic, cervical or axillary region and overlap of fields with current treatment
* OR life expectancy of less than 2 years
* OR pre-existing conditions or comorbidities making toxicity evaluation difficult, e.g. skin disorders
* OR pregnant or breast feeding
* OR mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* OR patient unlikely to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Breast retraction | 2 years after radiotherapy
  Rate of breast retraction or volume loss after radiotherapy

SECONDARY OUTCOMES:
Acute toxicity - Dermatitis | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Dermatitis measured by CTCAE v4.03
Acute toxicity - Desquamation | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Desquamation measured by CTCAE v4.03
Acute toxicity - Breast oedema | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Breast oedema measured by CTCAE v4.03
Acute toxicity - Shoulder range of motion | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Shoulder range of motion measured by maximal excursion in abduction-adduction and anteversion-retroversion, in degrees from anatomical reference position
Acute toxicity - Arm circumference | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Arm circumference measured in cm 15 cm above and below medial epicondyle
Acute toxicity - Breast symptoms - pain | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Breast pain measured on a scale: 0 (no pain) - 1 (pain on contact) - 2 (pain on contact and also occasionally spontaneous) - 3 (pain on contact and regularly spontaneous) - 4 (pain medication needed and specify which)
Acute toxicity - Breast symptoms - sense of heaviness | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Sense of breast heaviness defined as present or absent.
Acute toxicity - Breast symptoms - itching | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Itching in the breast on a scale: 0 (no itching) - 1 (occasional itching) - 2 (regular itching)
Acute toxicity - Arm Symptoms - Pain | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Arm pain measured on a scale: 0 (no pain) - 1 (pain on contact) - 2 (pain on contact and also occasionally spontaneous) - 3 (pain on contact and regularly spontaneous) - 4 (pain medication needed and specify which)
Acute toxicity - Arm Symptoms - Sense of heaviness | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Sense of arm heaviness defined as present or absent.
Acute toxicity - Shoulder symptoms - Pain | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Pain in the irradiated shoulder as defined on a scale: 0 (no pain) - 1 (occasional pain) - 2 (regular pain)
Acute toxicity - Shoulder symptoms - Impaired shoulder mobility | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Impaired shoulder mobility on the irradiated side defined as present or absent
Acute toxicity - Pain not in arm/shoulder/breast | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Pain present in any other region than arm, shoulder or breast, defined on a scale: 0 (no pain) - 1 (occasional pain) - 2 (regular pain). Painful locations are indicated on a figure.
Acute toxicity - Dysphagia | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Dysphagia measured according to CTCAE v4.03
Acute toxicity - Dyspnea | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Dyspnea measured according to CTCAE v4.03
Acute toxicity - Cough | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Cough measured according to CTCAE v4.03
Acute toxicity - Cardiac toxicity | Baseline and from radiation initiation until 8-16 days after radiation treatment
  Troponin T value at last treatment session ± 1 day compared with baseline measurement.
Non-breast retraction late treatment related toxicity | Baseline and from 6 months post radiotherapy until 5 years after radiotherapy
  breast oedema, telangiectasia, color changes, fibrosis, shoulder symptoms, breast symptoms, arm symptoms, brachial plexopathy, heart toxicity, dyspnea, thyroid function, pain, fatigue.
Cosmesis | Baseline, 1st visit after radiotherapy and at year 1, 2 and 5
  Photographic image analysis using BCCT.core using frontal images with different arm positions. Reported cosmetic outcome is evaluated with radiotherapy specific items of the Breast Q questionnaire
Quality of life - General | At baseline and at 1, 2 and 5 years after radiotherapy
  EORTC questionnaire QLQ-C30
Quality of life - Breast specific questionnaire | At baseline and at 1, 2 and 5 years after radiotherapy
  Supplementing the general quality of life outcome (QLQ-C30) with breast specific questionnaire using the EORTC QLQ-BR23 tool
Locoregional and distant tumor control | At 1, 2 and 5 years after radiotherapy
  Locoregional and distant tumor control
Treatment duration | At 3 weeks
  Time registration from the moment the patient climbs the treatment couch until end of radiation. The first fraction is not measured as unforeseen problems in the workflow, questions or difficulties might delay treatment and falsify the results. The moment the patient mounts the treatment couch as well as the moment she climbs down, will be registered using a remote sensor. The beam on time is automatically registered by the treatment software.
Dose parameters of target tissues/organs at risk | After treatment planning (Week 1-2 after inclusion)
  Data extracted from dose-volume histograms (DVHs) and associated DVH planning files. the data are extracted from the developped treatment plan before treatment is initiated. Discrete values will be evaluated for all patients, more precisely the following:
  D02 as a surrogate for Dmax, D05, D50, D95, D100, mean dose. All these values are reported in Gray (Gy)
  Parameters evaluated for OARs:
  - Mean dose, D02, D05, all in Gray
Volume parameters of targets/organs at risk/hot spots - volume of the structures | After treatment planning (Week 1-2 after inclusion)
  Data extracted from dose-volume histograms (DVHs) and associated DVH planning files. the data are extracted from the developped treatment plan before treatment is initiated.
  Volume of the targets and organs at risk is measured in cubic centimeters (cm³). Hot spots are defined as regions receiving either 105 or 107 % of the prescribed dose or more.
Volume parameters of targets/organs at risk - relative volume receiving a certain dose | After treatment planning (Week 1-2 after inclusion)
  Data extracted from dose-volume histograms (DVHs) and associated DVH planning files. the data are extracted from the developped treatment plan before treatment is initiated.
  For Organs at risk, a V5, V10, V20, V30 will be calculated. This is the relative volume of a the structure receiving a dose of 5, 10, 20 or 30 Gy. The value is measured as a percentage (%) of the total structure volume.
Setup accuracy | Before each scheduled radiation treatment session (every treatment day starting from radiotherapy start until ± 3 weeks later)
  Cone beam computed tomography verification directly prior to each scheduled radiation treatment session to determine shift between planned positioning and actual positioning. Shifts are performed and registered in laterolateral, craniocaudal and anteroposterior directions. No rotations are performed.
Treatment cost | Baseline, 1st visit after radiotherapy and at year 1, 2 and 5
  Cost-Utility Analysis (CUA) using the EuroQoL 5D tool.

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Vandecasteele, MD, PhD, Principal Investigator — UZ Ghent
Locations (1):
- Radiotherapy department, UZ Ghent, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Mulliez T, Veldeman L, van Greveling A, Speleers B, Sadeghi S, Berwouts D, Decoster F, Vercauteren T, De Gersem W, Van den Broecke R, De Neve W. Hypofractionated whole breast irradiation for patients with large breasts: a randomized trial comparing prone and supine positions. Radiother Oncol. 2013 Aug;108(2):203-8. doi: 10.1016/j.radonc.2013.08.040. Epub 2013 Sep 14. PMID 24044803
- [Background] Kirby AM, Evans PM, Donovan EM, Convery HM, Haviland JS, Yarnold JR. Prone versus supine positioning for whole and partial-breast radiotherapy: a comparison of non-target tissue dosimetry. Radiother Oncol. 2010 Aug;96(2):178-84. doi: 10.1016/j.radonc.2010.05.014. Epub 2010 Jun 17. PMID 20561695
- [Background] Mulliez T, Van de Velde J, Veldeman L, De Gersem W, Vercauteren T, Speleers B, Degen H, Wouters J, Van Hoof T, van Greveling A, Monten C, Berwouts D, De Neve W. Deep inspiration breath hold in the prone position retracts the heart from the breast and internal mammary lymph node region. Radiother Oncol. 2015 Dec;117(3):473-6. doi: 10.1016/j.radonc.2015.09.030. Epub 2015 Oct 8. PMID 26455452
- [Background] Mulliez T, Veldeman L, Speleers B, Mahjoubi K, Remouchamps V, Van Greveling A, Gilsoul M, Berwouts D, Lievens Y, Van den Broecke R, De Neve W. Heart dose reduction by prone deep inspiration breath hold in left-sided breast irradiation. Radiother Oncol. 2015 Jan;114(1):79-84. doi: 10.1016/j.radonc.2014.11.038. Epub 2014 Dec 9. PMID 25497557
- [Background] Deseyne P, Speleers B, De Neve W, Boute B, Paelinck L, Van Hoof T, Van de Velde J, Van Greveling A, Monten C, Post G, Depypere H, Veldeman L. Whole breast and regional nodal irradiation in prone versus supine position in left sided breast cancer. Radiat Oncol. 2017 May 26;12(1):89. doi: 10.1186/s13014-017-0828-6. PMID 28549483
- [Background] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Background] Monten C, Lievens Y, Olteanu LAM, Paelinck L, Speleers B, Deseyne P, Van Den Broecke R, De Neve W, Veldeman L. Highly Accelerated Irradiation in 5 Fractions (HAI-5): Feasibility in Elderly Women With Early or Locally Advanced Breast Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):922-930. doi: 10.1016/j.ijrobp.2017.01.229. Epub 2017 Feb 1. PMID 28366576